CLINICAL TRIAL: NCT05995041
Title: Universal CAR T Cells for the Treatment of Acute Myeloid Leukemia
Brief Title: Universal CAR-T Cells Targeting AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-23004
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Universal CAR T; CD33, CD123, CD38, CLL-1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple universal CAR T cells to treat AML (Experimental)
  Interventions: Biological: CLL-1, CD33, CD38 and/or CD123-specific universal CAR- T cells

INTERVENTIONS:
Biological: CLL-1, CD33, CD38 and/or CD123-specific universal CAR- T cells — Infusion of CLL-1, CD33, CD38 and/or CD123-specific universal CAR- T cells

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of universal CAR T-cell products targeting CLL-1, CD33, CD38 and CD123 in patients with relapsed and refractory AML. The study also aims to learn more about the function of the universal CAR T cells and their persistency in AML patients.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a malignant disease characterized by the rapid growth of myeloblasts that grow in the bone marrow and interferes with the generation of normal blood cells.Over the past years, several groups have demonstrated that CLL1, CD33, CD38 and CD123 are potential AML targets. CLL-1 (C-type lectin-like molecule-1) is a transmembrane glycoprotein, which is overexpressed in leukemic stem cells but absent in normal hematopoietic stem cells, suggesting that CLL-1 can be a promising target for targeted AML therapy. Although CAR-T cells have shown impressive anti-leukemic effect in B cell disease, CAR-T treatment for AML has proven to be more difficult. One of the reasons is because AML patients often has highly suppressed bone marrow function, and it is often difficult to obtain good quality of T cells for CAR-T preparation. In addition, AML progression can be acute and rapid, which can outpace the CAR-T expansion, and the time-consuming CAR-T manufacture process makes it more difficult to treat AML with autologous source of T cells By using universal type of CAR-T cells, the product can be supplied off-the-shelf without being customized from individual patients. In addition, the immediate availability means that patients with short disease remission time under severe bone marrow suppression may get a chance to be treated with CAR-T cells to achieve disease remission. In addition, those patients who suffer from long-term immunosuppression due to tumor microenvironment or myelosuppressive chemotherapy would have the option of treatment with the universal CAR-T cells.

The purpose of this study is to assess the feasibility, safety and efficacy of several AML-specific universal CAR-T products. Another goal is to learn more about the function of the universal CAR T cells and their persistency in the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Confirmed expression of CLL-1, CD123, CD38 and/or CD33 in AML blasts by immuno-histochemical staining or flow cytometry.
3. Karnofsky performance status (KPS) score is higher than 80 and life expectancy > 3 months.
4. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, total bilirubin ≤ 2.0mg/dL.
5. Hgb≥80g/L.
6. No cell separation contraindications.
7. Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
2. Active bacterial, fungal or viral infection not controlled by adequate treatment.
3. Known HIV or active hepatitis C virus (HCV) infection.
4. Pregnant or nursing women may not participate.
5. Use of glucocorticoid for systemic therapy within one week prior to entering the trial.
6. Previous treatment with any gene therapy products.
7. The bone marrow AML burden (MRD) is above 50%.
8. Patients, in the opinion of investigators, may not be able to comply with the study.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion | 6 months
  Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Clinical response | 1 year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-Immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No